CLINICAL TRIAL: NCT06368544
Title: Effect of Early Gait Training on Knee Cartilage Degeneration After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M2023816
Record Dates: First submitted 2024-03-05; First posted 2024-04-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Injuries; Cartilage Degeneration
Keywords: anterior cruciate ligament injuries; gait training; Cartilage biochemical characteristics; anterior cruciate ligament reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait intervention group (Experimental): On the basis of routine standardized rehabilitation procedures, in Early gait intervention training under the condition of weight loss
  Interventions: Other: lower-body positive-pressure
- Standardized rehabilitation control group (No Intervention): Only standardized rehabilitation training

INTERVENTIONS:
Other: lower-body positive-pressure — By increasing the chamber in the lower body around Pressure acts as a counterweight to gravity
  Arms: Gait intervention group

SUMMARY:
A randomized controlled clinical study was conducted to elucidate the relationship between the lower extremity biomechanics of patients undergoing early gait training after ACLR surgery.The relationship between the biochemical characteristics of cartilage and the biomechanical risk index were proposed to providing exercise guidance and training for ACLR people and it is suggested that it can prevent and reduce the risk of cartilage degeneration early after operation.

DETAILED DESCRIPTION:
In this randomized controlled clinical study, patients with primary unilateral ACL rupture were included. In addition to standardized rehabilitation training content, gait training intervention under weight loss was added to the subjects in the early postoperative period. The control group only received standardized rehabilitation training. Based on motion testing and dynamic analysis, the influence of early postoperative gait training on postoperative gait biomechanical characteristics was explored. And the influence of early cartilage health status; Based on functional MRI, the effects of early postoperative gait training on biochemical parameters of knee tibiofemoral and patellofemoral cartilage were investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACL rupture were diagnosed by MRI;
2. Unilateral ACL rupture for the first time should be performed in our hospital (Department of Sports Medicine, Peking University Third Hospital)The art of reconstruction;
3. Normal BMI range: 18.5-23.9 kg/m2;
4. Within 6 months from the trauma;
5. The affected knee joint has passed the acute stage, no obvious redness, pain,inflammation, and limited joint motion,basically restore joint motion.

Exclusion Criteria:

1. BMI<18.5 kg/m2 or BMI≥24 kg/m2);
2. There is a history of contralateral lower limb musculoskeletal system injury and surgery;
3. ACL injury time > 6 months;
4. Outerbridge damage rating Ⅲ and Ⅳ;
5. Patients with meniscal tears who are expected to undergo meniscal suture surgery at the time of ACLR surgery;
6. Serious injury to the posterior cruciate ligament, medial collateral ligament, or lateral collateral ligament;
7. There is metabolic syndrome (obesity, dyslipidemia, diabetes, etc.), which will involve articular cartilage Epidemic diseases, serious cardiovascular and cerebrovascular diseases, etc.;
8. Those who do not want to accept this treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait biomechanical data | from 3 months to 2 years
  Hip, knee and ankle joint angles and moments at the moment of landing and peak ground reaction force.
Gait biomechanical data | from 3 months to 2 years
  The maximum three-dimensional torque of the hip, knee and ankle during the support phase.
Gait biomechanical data | from 3 months to 2 years
  The maximum three-dimensional Angle and range of motion of the hip, knee and ankle joints during the whole gait cycle.
Gait biomechanical data | from 3 months to 2 years
  The symmetry index of Angle and torque of each joint.
Gait biomechanical data | from 3 months to 2 years
  The two groups of joint biomechanics and their gait touch information characteristics
Biochemical characteristics of knee cartilage | from 3 months to 2 years
  T1rho values of different regions of knee cartilage
Biochemical characteristics of knee cartilage | from 3 months to 2 years
  T2 mapping values of different regions of knee cartilage

CONTACTS AND LOCATIONS:
Overall Officials: ren shuang, doctor, Study Chair — Be affiliated with the organization
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided